CLINICAL TRIAL: NCT03475004
Title: Phase II Study of Pembrolizumab in Combination With Binimetinib and Bevacizumab in Patients With Refractory Colorectal Cancer
Brief Title: Study of Pembrolizumab, Binimetinib, and Bevacizumab in Patients With Refractory Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-0466.cc
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: Pembrolizumab; Binimetinib; Bevacizumab; Combination Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab; Bevacizumab; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety run-in (Other): Ten patients will be accrued to stage 1 and treated with standard doses of pembrolizumab, binimetinib and bevacizumab. If the standard doses are not tolerable and 2 or more patients experience a DLT, then patients would be enrolled in dose level -1 which would comprise of standard doses of pembrolizumab and bevacizumab but binimetinib would be at a dose lower of 30 mg PO BID. If 2 or more patients experience a DLT at dose level -1, then patients will be enrolled in dose level -2 which will comprise of standard doses of pembrolizumab and bevacizumab but a lower dose of binimetinib at 15 mg BID. Upon determination of the safety and tolerability of the treatment regimen, the study will proceed to stage 2.
  Interventions: Drug: Pembrolizumab; Drug: Bevacizumab; Drug: Binimetinib
- Cohort A (Experimental): Patients will start with 7-day run-in of binimetinib on day -7 of cycle 1 only. Pembrolizumab and bevacizumab will then be added to binimetinib on cycle 1 day +1. Cycle 1 will end on day 21. Patients will start treatment with pembrolizumab, binimetinib, and bevacizumab on day 1 of all subsequent cycles.
  Interventions: Drug: Pembrolizumab; Drug: Bevacizumab; Drug: Binimetinib
- Cohort B (Experimental): Patients will be treated with pembrolizumab, bevacizumab, and binimetinib together on day 1 of all cycles including cycle 1. Patients will start treatment with pembrolizumab, binimetinib, and bevacizumab on day 1 of all subsequent cycles.
  Interventions: Drug: Pembrolizumab; Drug: Bevacizumab; Drug: Binimetinib

INTERVENTIONS:
Drug: Pembrolizumab — An intravenous, potent and highly selective humanized monoclonal antibody of the immunoglobulin G4 (IgG4)/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda
Drug: Bevacizumab — The pharmacokinetics of bevacizumab are characterized by a slow CL, long half-life, and a volume of distribution consistent with limited extravascular distribution.
  Other Names: Avastin
Drug: Binimetinib — Binimetinib (MEK162/ARRY-438162) is an orally bioavailable, small molecule selective and potent mitogen-activated protein kinase (MEK) 1 and MEK 2 inhibitor.

SUMMARY:
This is an open-label, single-center, single-arm phase II clinical trial evaluating the combination of pembrolizumab, binimetinib, and bevacizumab in patients with metastatic colorectal adenocarcinoma who have not responded to prior therapy.

DETAILED DESCRIPTION:
This study will be done in two stages. In stage 1, ten patients will be treated with standard doses of pembrolizumab, binimetinib, and bevacizumab to ensure that the doses are safe and tolerable. In stage 2, patients will be enrolled into either cohort A, where they will be treated with a 7-day run-in of binimetinib, followed by pembrolizumab, bevacizumab, and binimetinib combination treatment in 21 day cycles, or they will be enrolled to cohort B, which does not include the 7-day run-in of binimetinib. Treatment in cohort B will include combination therapy of pembrolizumab, binimetinib, and bevacizumab from first day of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Age ≥ 18 years.
3. Able to comply with the study protocol, in the investigator's judgment.
4. Patient must state willingness to undergo pre- and post-treatment biopsies. According to the investigator's judgement, the planned biopsies should not expose the patient to substantially increased risk of complications.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or one.
6. Histologically confirmed unresectable metastatic colorectal adenocarcinoma.
7. Progression on at least two prior lines of therapy for unresectable metastatic colorectal adenocarcinoma.

   o Administration of bevacizumab previously does not impact study inclusion.
8. Measurable disease, according to RECIST v1.1. Note that lesions intended to be biopsied should not be target lesions.
9. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to first dose of study drug treatment:

   * WBC ≥ 2.5 and ≤ 15.0 × 109/L
   * ANC ≥ 1.5 × 109/L
   * Platelet count ≥ 100 × 109/L
   * Hemoglobin ≥ 9 g/dL without transfusion in the previous week
   * Albumin ≥ 2.5 g/dL
   * Serum bilirubin ≤ 1.5 x the upper limit of normal (ULN); patients with known Gilbert's disease may have a bilirubin ≤ 3.0 ×ULN
   * INR and PTT ≤ 1.5 × ULN; amylase and lipase ≤ 1.5 × ULN
   * AST, ALT, and alkaline phosphatase (ALP) ≤ 3 × ULN with the following exceptions:

     * Patients with documented liver metastases: AST and/or ALT ≤ 5 ×ULN
     * Patients with documented liver or bone metastases: ALP ≤ 5×ULN
   * Creatinine clearance ≥ 50 mL/min
10. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use of contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 180 days after the last study treatment. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
11. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 180 days after the last dose of study treatment. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Cancer-related exclusion criteria:

* Patients with known MSI-high status or unknown MSI status are not eligible for study entry.
* Patients with BRAF V600E mutations are not eligible for the study.
* Surgical procedure (surgical resection, wound revision or any other major surgery) or significant traumatic injury within 60 days prior to enrollment, or anticipation of need for major surgical procedure during the course of the study. Minor surgical procedure within 7 days (including placement of a vascular access device) of study Cycle 1 Day 1.

  1. Study-related biopsies are NOT considered surgical procedures under the exclusion criteria
* Untreated CNS metastases. Treatment of brain metastases, either by surgical or radiation techniques, must have been completed at least 4 weeks prior to initiation of study treatment.
* Treatment with any investigational agent or approved therapy within 21 days (Cycle 1 Day 1).
* Malignancies other than CRC within 3 years prior to Cycle 1 Day 1 with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year overall survival > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).
* Prior radiation therapy within 14 days prior to study Cycle 1 Day 1 and/or persistence of radiation-related adverse effects. However, palliative radiation therapy (as long as it does not involve target lesions) is permitted on the study.
* Prior allogeneic bone marrow transplantation or solid organ transplant for another malignancy in the past.
* Spinal cord compression not definitively treated with surgery and/or radiation.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
* Uncontrolled tumor related pain. Patients who require narcotic pain medication during screening should be on a stable dose regimen prior to Cycle 1 Day 1.

  2. Exclusion criteria related to study medication:
* Current or recent (within 10 days of study enrollment) use of acetylsalicylic acid (> 325 mg/day), clopidogrel (> 75 mg/day) or current or recent (within 10 days of first dose of bevacizumab) use of therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purpose. Note: The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks at the time of Cycle 1 Day 1. Prophylactic use of anticoagulants is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells, any components of Binimetinib, Pembrolizumab, or bevacizumab formulations or any premedications.
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD-1, anti-PD L1, anti-PD-L2 or MAPK pathway inhibitors (eg; BRAF, MEK, ERK inhibitors).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to randomization.

  3. Exclusion criteria based on autoimmune conditions:
* History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* History of non-infectious pneumonitis that required steroids or has current pneumonitis.
* Has an autoimmune disease that has required systemic treatment in the past 2 years with use of disease modifying agents, corticosteroids, or immunosuppressive drugs. Replacement therapy (eg; thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.

  4. Exclusion criteria based on organ function or medical history:
* History of clinically significant cardiac or pulmonary dysfunction including the following:

  1. Inadequately controlled hypertension (that is defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg that is treated or untreated).
  2. History of myocardial infarction within 6 months prior to first dose of study drug in Cycle.
  3. Prior history of hypertensive crisis or hypertensive encephalopathy.
  4. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, evidence of active pneumonitis on screening chest CT scan or non-infectious pneumonitis requiring steroids.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of Cycle 1 Day 1.
* History of stroke or transient ischemic attack within 6 months prior to Cycle 1 Day 1.
* Serious non-healing wound, active ulcer or untreated bone fracture.
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Cycle 1 Day 1.
* History of hemoptysis (≥one teaspoon of bright red blood per episode), or any other serious hemorrhage or at risk of bleeding (gastrointestinal history of bleeds, gastrointestinal ulcers, etc.). INR> 1.5 and aPTT > 1.5 × ULN within 7 days prior to Cycle 1 Day 1. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding.
* Life expectancy of < 12 weeks.
* Any previous venous thromboembolism≥ Grade 3.
* Proteinuria at screening as demonstrated by urine dipstick ≥ 2+ or 24-hour. proteinuria > 1.0 g.
* Left ventricular ejection fraction (LVEF) below institutional lower limit of normal.
* Uncontrolled serious medical or psychiatric illness.
* Pregnant or lactating, or intending to become pregnant during the study. Women who are not post-menopausal (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) or surgically sterile must have a negative serum pregnancy test within 14 days prior to Cycle 1 Day 1.

  5. Ocular exclusion criteria:
* History or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy, retinal vein occlusion or neovascular macular degeneration.
* Patients will be excluded if they have the following risk factors for retinal vein occlusion: Uncontrolled glaucoma with intraocular pressure ≥21 mmHg. Serum cholesterol ≥ Grade 2. Hypertriglyceridemia ≥ Grade 2. Hyperglycemia (fasting) ≥ Grade 2

  6. Exclusion criteria based on infectious diseases:
* Active infection requiring IV antibiotics at screening.
* Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening). Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to Cycle 1 Day 1.
* Patients with active hepatitis C. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Known HIV infection.
* Influenza vaccination should be given during influenza season. Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1 Day 1 or at any time during the study and for at least 5 months after the last dose of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2024-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lieu, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Universtiy of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Other: Safety run-in: Ten patients will be accrued to stage 1 and treated with standard doses of pembrolizumab, binimetinib and bevacizumab. If the standard doses are not tolerable and 2 or more patients experience a DLT, then patients would be enrolled in dose level -1 which would comprise of standard doses of pembrolizumab and bevacizumab but binimetinib would be at a dose lower of 30 mg PO BID. If 2 or more patients experience a DLT at dose level-1, then patients will be enrolled in dose level -2 which will comprise of standard doses of pembrolizumab and bevacizumab but a lower dose of binimetinib at 15 mg BID. Upon determination of the safety and tolerability of the treatment regimen, the study will proceed to stage 2.
- Experimental: Cohort A: Patients will start with 7-day run-in of binimetinib on day -7 of cycle 1 only. Pembrolizumab and bevacizumab will then be added to binimetinib on cycle 1 day +1. Cycle 1 will end on day 21. Patients will start treatment with pembrolizumab, binimetinib, and bevacizumab on day 1 of all subsequent cycles.
- Experimental: Cohort B: Patients will be treated with pembrolizumab, bevacizumab, and binimetinib together on day 1 of all cycles including cycle 1. Patients will start treatment with pembrolizumab, binimetinib, and bevacizumab on day 1 of all subsequent cycles.
Period: Overall Study
Arm/Group | Other: Safety run-in | Experimental: Cohort A | Experimental: Cohort B
Started | 11 | 21 | 21
Completed | 10 | 20 | 20
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Safety run-in: Ten patients will be accrued to stage 1 and treated with standard doses of pembrolizumab, binimetinib and bevacizumab. If the standard doses are not tolerable and 2 or more patients experience a DLT, then patients would be enrolled in dose level -1 which would comprise of standard doses of pembrolizumab and bevacizumab but binimetinib would be at a dose lower of 30 mg PO BID. If 2 or more patients experience a DLT at dose level-1, then patients will be enrolled in dose level -2 which will comprise of standard doses of pembrolizumab and bevacizumab but a lower dose of binimetinib at 15 mg BID. Upon determination of the safety and tolerability of the treatment regimen, the study will proceed to stage 2.
- Total: Total of all reporting groups
Arm/Group | Safety run-in | Cohort A | Cohort B | Total
Number analyzed (Participants) | 11 | 21 | 21 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 16 | 20 | 43
  >=65 years | 4 | 5 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11.4) | 52 (13.1) | 53 (9.8) | 53.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 7 | 26
  Male | 6 | 7 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 19 | 21 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 7 | 18 | 18 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 11 | 21 | 21 | 53

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Each study subject will be considered as a responder if their best CT imaging result is either CR (complete response) or PR (partial response) based on the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) evaluation criteria.
Time Frame: Study beginning to study end; 12 months
Population: All eligible subjects with response data
Measure: Count of Participants; unit: Participants
Groups:
- Safety Run-In: Phase 1: Triplet tx w/o run-in of binimetinib (see 'Arms and Interventions' description in Protocol Section)
- Cohort A: Phase 2: Triplex tx with 7-day run-in of binimetinib (see 'Arms and Interventions' in Protocol Section)
- Cohort B: Phase 2: Triplex tx w/o 7-day run-in of binimetinib (see 'Arms and Interventions' of Protocol Section)
Arm/Group | Safety Run-In | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 18 | 18
Participants | 1 | 3 | 2

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: The median progression-free survival was calculated using the Kaplan-Meier product-limit method.
Time Frame: Study start date to first sign of disease progression or death, whichever comes first.
Population: All patients who had follow-up data. Among the 50 total subjects, subjects 11, 19, 32, 33, and 53 did not have follow-up data. This resulted in 45 subjects being included in the PFS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Safety Run-In: Phase 1: Triplet tx w/o run=in of binimetinib (see 'Arms and Interventions' of Protocol Section)
- Cohort A: Phase 2: Triplet tx w/ 7-day run-in of binimetinib (see 'Arms and Interventions' of Protocol Section)
- Cohort B: Phase 2: Triplet tx w/o 7-day run-in of binimetinib (see 'Arms and Interventions' of Protocol Section)
Arm/Group | Safety Run-In | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 18 | 18
Months | 8.7 [2.2 to NA] — The upper limit of this 95% CI is infinity (and the entry 'Infinity' cannot be made) | 7.6 [2.8 to NA] — The upper limit of this 95% CI is infinity (and the entry 'Infinity' cannot be made) | 5.8 [2.8 to 6.9]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time (measured in months) from each subject starting treatment until either death (from any cause) or being censored at their last contact.
Time Frame: Time (measured in months) from each subject starting treatment until either death (from any cause) or being censored at their last contact.
Population: All 50 subjects enrolled onto the trial.
Measure: Median (95% Confidence Interval); unit: Months-to-Death
Groups:
- Safety Run-In: Phase 1: Triplet tx w/o run-in of binimetinib (see 'Arms and Interventions' of Protocol Section)
Arm/Group | Safety Run-In | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 20 | 20
Months-to-Death | 12.6 [1.9 to 20.7] | 9.3 [4.5 to NA] — The upper limit of this 95% CI is infinity (and the entry 'Infinity' cannot be made) | 8.5 [5.9 to 10.7]

4. Secondary Outcome: Adverse Events
Description: Grade 1, 2, 3, 4, or 5 adverse events (AE) as defined by CTCAE v4 were summarized. All adverse events summarized were non-baseline AEs (i.e. each AE was not present at baseline). AEs were summarized by generating counts of AEs by AE description and severity, but no formal statistical test was performed on the AEs.
  For the purpose of this section, the outcome measure will be defined as the number of subjects who had at least 1 AE.
Time Frame: Study beginning to study end, 12 months
Population: Adverse events from all subjects were evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Phase 2: Triplet tx w 7-day run-in of binimetinib (see 'Arms and Interventions' of Protocol Section)
- Cohort B: Phase 2: Triplet tx w/o 7-day run-in of binimetinib (see 'Arms and Interventions' of Protocol Section
Arm/Group | Safety Run-In | Cohort A | Cohort B
Number analyzed (Participants) | 10 | 20 | 20
Participants | 10 | 20 | 20

ADVERSE EVENTS:
Time Frame: 3 years, 4 months
Arm/Group | Safety run-in | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/11 | 4/21 | 1/21
Serious Adverse Events (participants affected / at risk) | 3/11 | 11/21 | 8/21
Other Adverse Events (participants affected / at risk) | 11/11 | 21/21 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety run-in (N=11) | Cohort A (N=21) | Cohort B (N=21)
Dehydration (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Leg Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Colon Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
alanine aminotransferase increase (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (General disorders) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 4 (4) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (General disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety run-in (N=11) | Cohort A (N=21) | Cohort B (N=21)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
CPK Increased (Blood and lymphatic system disorders) | 7 (9) | 5 (8) | 1 (1)
Dehydration (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 8 (10) | 17 (40) | 15 (19)
Alkaline Phosphatase Increased (Blood and lymphatic system disorders) | 2 (2) | 5 (6) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 1 (1)
Lipase Increased (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (2)
Oral Mucositis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 9 (16) | 10 (15) | 11 (16)
Nausea (General disorders) | 8 (9) | 8 (9) | 7 (10)
Alanine Aminotransferase Increase (Blood and lymphatic system disorders) | 2 (2) | 4 (7) | 3 (3)
Aspartate Aminotransferase Increase (Blood and lymphatic system disorders) | 2 (3) | 6 (13) | 3 (4)
Hypertension (Blood and lymphatic system disorders) | 6 (11) | 7 (10) | 4 (4)
Ejection Fraction Decreased (Cardiac disorders) | 2 (2) | 3 (5) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0)
Platelet Count Decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Edema (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) | 9 (9)
Abdominal Pain (General disorders) | 3 (3) | 8 (9) | 9 (9)
Retinopathy (Eye disorders) | 5 (6) | 1 (1) | 1 (1)
Blurred Vision (Eye disorders) | 1 (2) | 3 (3) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 2 (2) | 1 (1)
Vomiting (General disorders) | 4 (5) | 4 (4) | 1 (2)
Proteinuria (Renal and urinary disorders) | 3 (4) | 6 (12) | 6 (8)
Colitis (Gastrointestinal disorders) | 1 (2) | 2 (3) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (8) | 10 (12) | 15 (18)
Back Pain (General disorders) | 4 (4) | 6 (9) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 4 (4) | 3 (4)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (2) | 4 (5)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 2 (3)
Hot Flashes (General disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Papulopustular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 2 (3) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 5 (5) | 5 (5)
Anorexia (General disorders) | 1 (1) | 1 (1) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Confusion (General disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0) | 1 (2)
Dysarthria (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Anal Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asystole (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Melena (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Increased Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated Cholesterol (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 6 (6) | 5 (6)
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Ear Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Disorders (Eye disorders) | 1 (1) | 3 (3) | 1 (1)
Flank Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (5) | 1 (1) | 2 (4)
General Disorders (General disorders) | 1 (1) | 3 (13) | 3 (6)
Muscle weakness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Hypertriglyceridemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 1 (1) | 2 (2) | 1 (1)
Intestinal stoma site bleeding (General disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory Impairment (General disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7) | 4 (4)
Neck pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PTSD (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal anastomotic leak (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (General disorders) | 2 (2) | 0 (0) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Vaginal Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachments (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Seizure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Serum amylase increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sore throat (General disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vaginal Inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular Disorder (clot) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Vasovagal reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Watering Eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperlipidemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03475004/Prot_SAP_ICF_000.pdf